CLINICAL TRIAL: NCT01728844
Title: A Randomized, Double-Blind, Controlled, Multicenter Dose Verification Clinical Trial to Evaluate the Safety and Effectiveness of GUIDOR® Growth Factor Enhanced Bone Graft Substitute for the Treatment of Periodontal Defects 6-months Post-Surgery
Brief Title: GUIDOR® Growth Factor Enhanced Bone Graft Substitute for the Treatment of Periodontal Defects 6-months Post-Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunstar Americas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLP-2011-10-31-1
Record Dates: First submitted 2012-11-01; First posted 2012-11-20 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-08

CONDITIONS: Alveolar Bone Loss; Periodontal Diseases
Keywords: bone grafting; alveolar bone loss; periodontal diseases
MeSH Terms: conditions — Alveolar Bone Loss; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- beta-tricalcium phosphate alone (Active Comparator): beta-tricalcium phosphate alone
  Interventions: Device: beta-tricalcium phosphate alone
- GFeBGS 0.1% (Experimental): GFeBGS consisting of beta-tricalcium phosphate + 0.1% recombinant human basic fibroblast growth factor (rh-bFGF)
  Interventions: Device: GFeBGS 0.1%
- GFeBGS 0.3% (Experimental): GFeBGS consisting of beta-tricalcium phosphate + 0.3% rh-bFGF
  Interventions: Device: GFeBGS 0.3%
- GFeGBS 0.4% (Experimental): GFeBGS consisting of beta-tricalcium phosphate + 0.4% rh-bFGF
  Interventions: Device: GFeBGS 0.4%

INTERVENTIONS:
Device: beta-tricalcium phosphate alone
  Arms: beta-tricalcium phosphate alone
Device: GFeBGS 0.1%
  Arms: GFeBGS 0.1%
Device: GFeBGS 0.3%
  Arms: GFeBGS 0.3%
Device: GFeBGS 0.4%
  Arms: GFeGBS 0.4%

SUMMARY:
GUIDOR Growth Factor Enchanted Bone Graft Substitute (GFeBGS) when used in periodontal surgery will shown greater gum and bone regeneration when compare to bone graft substitute alone. Also, to find the optimal dose.

DETAILED DESCRIPTION:
This will be a prospective, randomized, double-blinded, controlled, multi-center, dose-verification clinical study in subjects who require surgical intervention to treat a qualifying periodontal defect.

Subjects 25 years and older with advanced periodontal disease in at least one site requiring surgical treatment to correct a bone defect.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age of 25 and older
* Must have read, understood, and signed a consent form
* Must be able and willing to follow study procedures and instructions
* Must have undergone thorough scaling and root planing of the target tooth and be expected to demonstrate good plaque control after instruction in oral hygiene
* The target tooth must exhibit the following:

  * A pocket depth of 7 mm or greater
  * After surgical debridement, 4 mm or greater intrabony defect with at least 1 bony wall
  * Sufficient keratinized tissue to allow complete tissue coverage of the defect
  * Radiographic base of defect at least 3 mm coronal to the apex of the tooth

Exclusion Criteria:

* Failure to maintain adequate oral hygiene during the screening phase
* Women of child-bearing potential
* A history within the last 6 months of HIV, Type IV heart disease, or end-stage renal disease
* A history of oral cancer or any other cancer (exception: subjects with a history of skin cancers such as squamous and basal carcinoma with end of treatment at least 6 months ago and/or prostate cancer with end of treatment at least 5 years ago may be enrolled)
* A history within 12 months of previous open flap periodontal surgery on the study tooth.
* A diagnosis of pre-malignant oral lesion(s)
* A traumatic occlusion of the target tooth
* Target "study" tooth exhibiting Grade III mobility
* Maxillary molars or maxillary first premolar with a prominent mesial concavity
* Study tooth exhibiting a Class II or greater furcation defect
* Clinical or radiographic signs of untreated acute or chronic periapical infection at the surgical site, apical pathology, root fracture, severe root irregularities, cemental pearls, cervical enamel projections not easily removed by odontoplasty, untreated carious lesions at the cemento-enamel junction (CEJ) or on the root surface, or restorations with open or otherwise defective margins at or below the CEJ
* A history within the last 6 months of the daily use of any tobacco products besides cigarettes (smokeless chewing tobacco, pipe or cigar smoking), or of smoking more than 10 cigarettes per day
* Subjects participating in other clinical trials within 30 days of enrollment
* Subjects having uncontrolled endocrine-induced diseases (e.g. uncontrolled diabetes mellitus and hyperparathyroidism)
* Subjects undergoing current therapy with systemic steroids or other drugs that significantly alter bone metabolism
* Subjects with Localized Juvenile Periodontitis (LJP) sites in the oral cavity

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L. Cochran, DDS, PhD, Principal Investigator — University of Texas Health Sciences Center at San Antonio
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Regenerative Solutions, Fullerton, California
  - Drs. McClain and Schallhorn, Aurora, Colorado
  - University of Michigan, Ann Arbor, Michigan
  - Perio Health Professionals, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Cochran DL, Oh TJ, Mills MP, Clem DS, McClain PK, Schallhorn RA, McGuire MK, Scheyer ET, Giannobile WV, Reddy MS, Abou-Arraj RV, Vassilopoulos PJ, Genco RJ, Geurs NC, Takemura A. A Randomized Clinical Trial Evaluating rh-FGF-2/beta-TCP in Periodontal Defects. J Dent Res. 2016 May;95(5):523-30. doi: 10.1177/0022034516632497. Epub 2016 Feb 23. PMID 26908630

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled at 6 dental clinical centers between November 2012 and December 2013.
Groups:
- Beta-tricalcium Phosphate Alone: beta-tricalcium phosphate + placebo vehicle
Period: Overall Study
Arm/Group | Beta-tricalcium Phosphate Alone | GFeBGS 0.1% | GFeBGS 0.3% | GFeGBS 0.4%
Started | 22 | 21 | 22 | 23
Completed | 21 | 21 | 22 | 21
Not Completed | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beta-tricalcium Phosphate Alone | GFeBGS 0.1% | GFeBGS 0.3% | GFeGBS 0.4% | Total
Number analyzed (Participants) | 22 | 21 | 22 | 23 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (10.7) | 59.7 (12.1) | 54.0 (10.6) | 54.0 (10.5) | 56.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 9 | 9 | 34
  Male | 13 | 14 | 13 | 14 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 3 | 1 | 10
  Not Hispanic or Latino | 21 | 16 | 19 | 22 | 78
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 3 | 2 | 2 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 4 | 3 | 11
  White | 16 | 15 | 14 | 18 | 63
  More than one race | 0 | 2 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Smoking history [Count of Participants; unit: Participants]
  Current smoker or smoked within past 6 months | 3 | 3 | 4 | 3 | 13
  Non-smoker | 19 | 18 | 18 | 20 | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Met the Success Criteria of Radiographic and Clinical Measurements
Description: The primary effectiveness endpoint is a composite endpoint that considers radiographic and clinical measurements at six months post-implantation: the amount of linear bone growth (LBG), which is assessed with the use of radiographs, and the regain from baseline of clinical attachment level (∆CAL), which is assessed clinically. Linear bone growth (LBG) in a vertical and horizontal direction is determined radiographically at six months post-implantation. The clinical attachment level (CAL) is the distance from the cemento-enamel junction (CEJ) (or other fixed reference point) generally along the long axis of the tooth to the deepest extent of the periodontal pocket. The success criteria are ΔCAL ≥1.5 mm and LBG ≥1 mm at 6 months after the treatment. Both the ∆CAL and LBG must meet the success criteria for a subject to be considered a success.
Time Frame: 6 months post-surgery
Population: The modified Intent-to-Treat population consisted of 83 subjects after two subjects were removed for lack of compliance with the study protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Beta-tricalcium Phosphate Alone | GFeBGS 0.1% | GFeBGS 0.3% | GFeGBS 0.4%
Number analyzed (Participants) | 20 | 21 | 21 | 21
Participants | 16 | 15 | 19 | 17

2. Secondary Outcome: Change in Clinical Attachment Level at 3 Months
Description: The clinical attachment level is the distance from the cemento-enamel junction (or other fixed reference point) generally along the long axis of the tooth to the deepest extent of the periodontal pocket. Change = (3 months measurement - Baseline measurement)
Time Frame: Baseline and 3 months post-surgery
Population: The modified Intent-to-Treat population consisted of 84 subjects after a subject was removed for lack of compliance with the study protocol.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Beta-tricalcium Phosphate Alone | GFeBGS 0.1% | GFeBGS 0.3% | GFeGBS 0.4%
Number analyzed (Participants) | 20 | 21 | 21 | 22
mm | 3.1 (1.4) | 2.9 (1.7) | 3.1 (1.6) | 3.5 (1.7)

3. Secondary Outcome: Change in Clinical Attachment Level at 6 Months
Description: The clinical attachment level is the distance from the cemento-enamel junction (or other fixed reference point) generally along the long axis of the tooth to the deepest extent of the periodontal pocket. Change = (6 months measurement - Baseline measurement)
Time Frame: Baseline and 6 months post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Beta-tricalcium Phosphate Alone | GFeBGS 0.1% | GFeBGS 0.3% | GFeGBS 0.4%
Number analyzed (Participants) | 20 | 21 | 21 | 21
mm | 2.9 (2.1) | 2.5 (2.1) | 3.0 (1.4) | 3.6 (1.8)

4. Secondary Outcome: Linear Bone Growth at 6 Months
Description: Linear measurement of bone height in millimeters along mesial and/or distal root surfaces of the defect site is captured radiographically at baseline and 6 months. Linear Bone Growth = (Baseline measurement - 6 months measurement)
Time Frame: Baseline and 6 months post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Beta-tricalcium Phosphate Alone | GFeBGS 0.1% | GFeBGS 0.3% | GFeGBS 0.4%
Number analyzed (Participants) | 20 | 21 | 21 | 21
mm | 3.1 (1.8) | 3.0 (1.2) | 3.7 (1.3) | 3.6 (2.1)

5. Secondary Outcome: Percent Bone Fill at 6 Months
Description: Linear measurement of bone height in millimeters along mesial and/or distal root surfaces of the defect site is captured radiographically at baseline and 6 months. Percent Bone Fill is calculated by dividing Linear Bone Growth at 6 months by bone height at baseline.
Time Frame: Baseline and 6 months post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of bone height change
Arm/Group | Beta-tricalcium Phosphate Alone | GFeBGS 0.1% | GFeBGS 0.3% | GFeGBS 0.4%
Number analyzed (Participants) | 20 | 21 | 21 | 21
percentage of bone height change | 62.5 (26.4) | 61.0 (23.0) | 74.6 (20) | 71.1 (37.8)

6. Secondary Outcome: Pocket Depth Change at 3 Months
Description: Length from free gingival margin to the base of the pocket in millimeter is measured with North Carolina 15 mm periodontal probes. Pocket Depth Change = (3 months measurement - Baseline measurement)
Time Frame: Baseline and 3 months post-surgery
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Beta-tricalcium Phosphate Alone | GFeBGS 0.1% | GFeBGS 0.3% | GFeGBS 0.4%
Number analyzed (Participants) | 20 | 21 | 21 | 22
mm | 3.7 (1.4) | 3.5 (1.4) | 3.5 (1.6) | 3.8 (1.1)

7. Secondary Outcome: Pocket Depth Change at 6 Months
Description: Length from free gingival margin to the base of the pocket in millimeter is measured with North Carolina 15 mm periodontal probes. Pocket Depth Change = (6 months measurement - Baseline measurement)
Time Frame: Baseline and 6 months post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Beta-tricalcium Phosphate Alone | GFeBGS 0.1% | GFeBGS 0.3% | GFeGBS 0.4%
Number analyzed (Participants) | 20 | 21 | 21 | 22
mm | 3.7 (1.2) | 2.9 (2.0) | 3.4 (1.0) | 3.7 (1.0)

8. Secondary Outcome: Change in Gingival Recession at 3 Months
Description: Length from the free gingival margin to the CEJ is measured in millimeter with North Carolina 15 mm periodontal probes. Gingival Recession = (3 months measurement - Baseline measurement)
Time Frame: Baseline and 3 months post-surgery
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Beta-tricalcium Phosphate Alone | GFeBGS 0.1% | GFeBGS 0.3% | GFeGBS 0.4%
Number analyzed (Participants) | 20 | 21 | 21 | 21
mm | -0.6 (1.4) | -0.6 (1.1) | -0.3 (1.2) | -0.3 (1.2)

9. Secondary Outcome: Change in Gingival Recession at 6 Months
Description: Length from the free gingival margin to the CEJ is measured in millimeter with North Carolina 15 mm periodontal probes. Gingival Recession = (6 months measurement - Baseline measurement)
Time Frame: Baseline and 6 months post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Beta-tricalcium Phosphate Alone | GFeBGS 0.1% | GFeBGS 0.3% | GFeGBS 0.4%
Number analyzed (Participants) | 20 | 21 | 21 | 21
mm | -0.7 (1.5) | -0.4 (1.0) | -0.4 (1.1) | -0.1 (1.3)

10. Post Hoc Outcome: Number of Participants That Met the Success Criteria of Radiographic and Clinical Measurements (Updated Success Criteria)
Description: The primary effectiveness endpoint is a composite endpoint that considers radiographic and clinical measurements at six months post-implantation: the amount of linear bone growth (LBG), which is assessed with the use of radiographs, and the regain from baseline of clinical attachment level (∆CAL), which is assessed clinically. Linear bone growth (LBG) in a vertical and horizontal direction is determined radiographically at six months post-implantation. The clinical attachment level (CAL) is the distance from the cemento-enamel junction (CEJ) (or other fixed reference point) generally along the long axis of the tooth to the deepest extent of the periodontal pocket. The updated success criteria are ΔCAL ≥1.5 mm and LBG ≥ 2.5 mm at 6 months after the treatment. Both the ∆CAL and LBG must meet the success criteria for a subject to be considered a success.
Time Frame: 6 months post-surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Beta-tricalcium Phosphate Alone | GFeBGS 0.1% | GFeBGS 0.3% | GFeGBS 0.4%
Number analyzed (Participants) | 20 | 21 | 21 | 21
Participants | 9 | 10 | 15 | 15

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Beta-tricalcium Phosphate Alone | GFeBGS 0.1% | GFeBGS 0.3% | GFeGBS 0.4%
All-Cause Mortality (participants affected / at risk) | 1/22 | 0/21 | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/22 | 1/21 | 1/22 | 0/23
Other Adverse Events (participants affected / at risk) | 4/22 | 6/21 | 2/22 | 10/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Beta-tricalcium Phosphate Alone (N=22) | GFeBGS 0.1% (N=21) | GFeBGS 0.3% (N=22) | GFeGBS 0.4% (N=23)
Bunion (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Basal cell carcinoma basal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 — Pre-existing condition was updated.
Chronic lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 — Pre-existing condition was updated.
Coma (Nervous system disorders) | 1 | 0 | 0 | 0 — An accident caused serious head trauma.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Beta-tricalcium Phosphate Alone (N=22) | GFeBGS 0.1% (N=21) | GFeBGS 0.3% (N=22) | GFeGBS 0.4% (N=23)
Application site pain (Injury, poisoning and procedural complications) | 0 | 4 | 2 | 5
Application site inflammation (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 5
Application site hyperaesthesia (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 0
Tooth abscess (Infections and infestations) | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution will submit the manuscript of the proposed publication to Sponsor at least 30 days prior to publication, and Sponsor shall have the right to review and comment upon the publication in order to protect Sponsor's confidential information. Upon Sponsor's written request, publication will be delayed up to 60 additional days to enable Sponsor to secure adequate intellectual property protection on Sponsor's intellectual property that would be affected by said publication.

DOCUMENTS (1):
  • Study Protocol (2013-02-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT01728844/Prot_000.pdf